CLINICAL TRIAL: NCT04404829
Title: The Effect of the Informational Manual Therapy for Improving Quiet Standing, Pain and Quality of Life in Healthy Individuals
Brief Title: Informational Manual Therapy to Improve Standing Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Rosa Cabanas Valdés, Universitat Internacional de Catalunya, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Poyet-Pialoux method
Record Dates: First submitted 2020-05-17; First posted 2020-05-28 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Balance Postural; Pain; Quality of Life
Keywords: balance; pain; quality of life; manual therapy
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The study has a one-group pretest-posttest design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Informational Manual Therapy (Experimental): It is an integral no orthopedic and very soft manual therapy
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — The first level of IMT was treated in this study: the objective is to harmonize the cranio-sacral and sacro-pelvic systems, as this is fundamental for maintaining good posture. The first therapeutic maneuvers should be focused on releasing of the sacrum and the pelvis. The first is considered a key area for the correct transmission of forces and loads from the lower limbs to the upper limbs and vice versa and shares the role of rigid elements for this purpose (bones) and tensile elements (muscles, ligaments, fascia) in the whole body. In this level. Compensatory injuries that the body has started after a primary injury are treated on this level, through the Fluidic Chains. The diagnosis of this level is performed by cranial somotopias. Practically all the treatment is carried out on the sacrum. The first step are the "fuses," which are vibration zones which act as a protection system for the body. These points sometimes stop working, which interrupts the correct movement of the PRM.
  Other Names: Poyet-Pialoux method

SUMMARY:
Objectives: The aim of this study is to assess the effect of Informational Manual Therapy (IMT) on quiet standing and quality of life in healthy individuals. The IMT also is known as the Poyet-Pialoux method, is a holistic, no orthopedic, and soft manual therapy.

Design: This is a one-group pretest-posttest design. It is a within-subjects experiment in which each participant is tested first under the control condition and then under the treatment condition.

Setting: University laboratory. Intervention: One IMT session was performed on 57 healthy individuals aged from 18 to 65 years. They were grouped into three age groups. The treatment session was performed by 5 therapists on two days. The primary outcome was quite standing assessed by the SATEL force platform. Secondary outcomes were bodily pain assessed by the pain sections of the 36-Item Short Form Survey (SF-36) and quality of life by EQ-5D-3L (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The primary outcome was evaluated before and immediately after treatment and after 7-10 days. The secondary outcomes were assessed after treatment and 3 weeks later.

DETAILED DESCRIPTION:
Methods Study Design: The study has a one-group pretest-posttest design. The personal data of individuals were kept confidential and the data were shared anonymously upon request from the principal researcher. The TREND statement will be followed.

Subjects Fifty-seven participants will be recruited to participate in this study; the sample was one of convenience. The inclusion and exclusion criteria are as follows: age from 18 to 65 years old, not having a positive diagnosis for any disease which influences balance, no participation in any other trial, not suffering from an injury in the 3 months before the study or fractures in the previous 6 months, and no falls in the previous month. All individuals provided informed consent before enrolment.

Intervention All the participants received a single session of 30-45 min of IMT. All the treatment sessions took place at the UIC laboratory. The IMT session was performed over two days by four physiotherapists and a doctor. All have more than five years of experience in IMT treatment.

The first level of IMT was treated in this study: the objective is to harmonize the Cranio-sacral and sacro-pelvic systems, as this is fundamental for maintaining good posture. The first therapeutic maneuvers should be focused on releasing of the sacrum and the pelvis. The first is considered a key area for the correct transmission of forces and loads from the lower limbs to the upper limbs and vice versa and shares the role of rigid elements for this purpose (bones) and tensile elements (muscles, ligaments, fascia) in the whole body. At this level. Compensatory injuries that the body has started after a primary injury are treated on this level, through the Fluidic Chains. This also includes the treatment of some traumatic injuries, such as cranial strains, the compression of spheno-basilar synchondrosis, injuries of the pelvis and occipital bone, and damage to the flexion-extension and lateral displacement of the vertebrae. The diagnosis of this level is performed by cranial somotopias (reflex points on the skull and face). Practically all the treatment is carried out on the sacrum. The first step is the "fuses," which are vibration zones that act as a protection system for the body (1). These points sometimes stop working, which interrupts the correct movement of the PRM: 1st fuse: Inn-trang (on the forehead between the two eyebrows, the 4th sacral vertebra is stimulated if it is not adjusted). A massage on the scalp in several very soft circles that goes from the frontal to the occipital area is performed 6 times. 2nd fuse: 1st dorsal vertebra, 4th cervical, 4th dorsal, and 3rd lumbar. 3rd fuse: C0 (base of the occipital), a zone of the 2nd sacral vertebra, and the space between the spines of the 2nd and 3rd dorsal vertebrae and finally point R1 (between the 2nd and 3 rd metatarsal). If any point is blocked it is treated and harmonized with a soft touch towards the occipital.

ELIGIBILITY:
Inclusion Criteria:

Healthy people

Exclusion Criteria:

Not having problems with balance, Not suffering from an injury in the 3 months before the study, Not suffering from a fracture in the previous 6 month before the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
static standing posture | baseline, pre-intervention
  It was assessed using the force platform Satel 40 Hz model PF2002, software v 33.5 8C (France).
static standing posture | immediately after the intervention
  It was assessed using the force platform Satel 40 Hz model PF2002, software v 33.5 8C (France).

SECONDARY OUTCOMES:
How much bodily pain have you had during the past 4 weeks? | baseline, pre-intervention
  by the 36-Item Short Form Survey (SF-36). 1 - None,2 - Very mild,3 - Mild, 4 - Moderate, 5 - Severe, - 6 very severe
How much bodily pain have you had during the past 4 weeks? | three weeks, post-intervention
  by the 36-Item Short Form Survey (SF-36). 1 - None,2 - Very mild,3 - Mild, 4 - Moderate, 5 - Severe, - 6 very severe
During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? | baseline, pre-intervention
  by the 36-Item Short Form Survey (SF-36). 1 - Not at all, 2 - A little bit, 3 - Moderately, 4 - Quite a bit, 5 - Extremely
During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? | three weeks after treatment
  by the 36-Item Short Form Survey (SF-36). 1 - Not at all, 2 - A little bit, 3 - Moderately, 4 - Quite a bit, 5 - Extremely
mobility | baseline, pre-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
mobility | three weeks post-intervention
  by the EQ-5D-3L questionnaire.Each dimension has 3 levels: no problems, some problems, and extreme problems
self-care | baseline, pre-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
self-care | three weeks post-intervention
  by the EQ-5D-3L questionnaire.Each dimension has 3 levels: no problems, some problems, and extreme problems
usual activities | baseline, pre-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
usual activities | three weeks post-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
pain/discomfort | baseline, pre-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
pain/discomfort | three weeks post-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
anxiety/depression | baseline, pre-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
anxiety/depression | three weeks post-intervention
  by the EQ-5D-3L questionnaire. Each dimension has 3 levels: no problems, some problems, and extreme problems
visual analogue scale for health | baseline, pre-intervention
  by the EQ-VAS, ranging from 0 ("worst possible") to 100 ("best possible").
visual analogue scale for health | three weeks post-intervention
  by the EQ-VAS, ranging from 0 ("worst possible") to 100 ("best possible").

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Cabanas Valdés, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
There is not any plan

REFERENCES:
- [Result] Bordoni B, Zanier E. Sutherland's legacy in the new millennium: the osteopathic cranial model and modern osteopathy. Adv Mind Body Med. 2015 Spring;29(2):15-21. PMID 25831430
- [Result] Tseui JJ. Eastern and western approaches to medicine. West J Med. 1978 Jun;128(6):551-7. PMID 664653
- [Result] Liem T, Neuhuber W. Osteopathic Treatment Approach to Psychoemotional Trauma by Means of Bifocal Integration. J Am Osteopath Assoc. 2020 Mar 1;120(3):180-189. doi: 10.7556/jaoa.2020.021. PMID 32091561
- [Result] Lee RP. The living matrix: a model for the primary respiratory mechanism. Explore (NY). 2008 Nov-Dec;4(6):374-8. doi: 10.1016/j.explore.2008.08.003. PMID 18984549
- [Result] Frymann VM. A study of the rhythmic motions of the living cranium. J Am Osteopath Assoc. 1971 May;70(9):928-45. No abstract available. PMID 5207590
- [Result] Ballester-Rodes M, Carreras-Costa F, Versyp-Ducaju T, Ballester-Rodes M, Mehta D. Field dynamics in atrioventricular activation. Clinical evidence of a specific field-to-protein interaction. Med Hypotheses. 2019 Mar;124:56-59. doi: 10.1016/j.mehy.2019.02.012. Epub 2019 Feb 2. PMID 30798917
- See also: Ostéopathie non structurelle ; à l'écoute du corps, une évolution de la méthode Poyet — https://halldulivre.com/livre/9782364031005-osteopathie-non-structurelle-a-l-ecoute-du-corps-une-evolution-de-la-methode-poyet-jean-marchandise-anne-paul-marchandise/